CLINICAL TRIAL: NCT02125461
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Multi-centre, International Study of MEDI4736 as Sequential Therapy in Patients With Locally Advanced, Unresectable Non-Small Cell Lung Cancer (Stage III) Who Have Not Progressed Following Definitive, Platinum-based, Concurrent Chemoradiation Therapy (PACIFIC)
Brief Title: A Global Study to Assess the Effects of MEDI4736 Following Concurrent Chemoradiation in Patients With Stage III Unresectable Non-Small Cell Lung Cancer
Acronym: PACIFIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4191C00001; 2014-000336-42 (EudraCT Number)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally advanced; Unresectable Non-Small Cell Lung Cancer; MEDI4736; PD-L1; Stage III Non-Small Cell Lung Cancer; Chemoradiation; Immune-mediated cancer therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI4736 (Experimental): MEDI4736 (intravenous infusion)
  Interventions: Drug: MEDI4736
- PLACEBO (Placebo Comparator): Placebo (matching placebo for intravenous infusion)
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 by intravenous infusion. Treatment from Day 1 for a maximum of 12 months or study drug withdrawal if this occurs earlier . The 2:1 ratio (MEDI4736 to placebo).
  Arms: MEDI4736
Other: PLACEBO — PLACEBO by intravenous infusion. Treatment from Day 1 for a maximum of 12 months or study drug withdrawal if this occurs earlier . The 2:1 ratio (MEDI4736 to placebo).
  Arms: PLACEBO

SUMMARY:
A Global Study to Assess the Effects of MEDI4736 following concurrent chemoradiation in Patients with Stage III Unresectable Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
A Phase III, Randomised, Double-blind, Placebo-controlled, Multi-centre, International Study of MEDI4736 as Sequential Therapy in Patients with Locally Advanced, Unresectable Non-Small Cell Lung Cancer (Stage III) Who Have Not Progressed Following Definitive, Platinum-based, Concurrent Chemoradiation Therapy (PACIFIC)

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years.
2. Documented evidence of NSCLC (locally advanced, unresectable, Stage III)
3. Patients must have received at least 2 cycles of platinum-based chemotherapy concurrent with radiation therapy.
4. World Health Organisation (WHO) Performance Status of 0 to 1.
5. Estimated life expectancy of more than 12 weeks.

Exclusion Criteria:

1. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody.
2. Active or prior autoimmune disease or history of immunodeficiency.
3. Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
4. Evidence of uncontrolled illness such as symptomatic congestive heart failure, uncontrolled hypertension or unstable angina pectoris.
5. Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy.
6. Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Dennis, MD, Study Director — AstraZeneca
Locations (204):
- United States (56):
  - Research Site, Chandler, Arizona
  - Research Site, Goodyear, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Oxnard, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Rosa, California
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Gordon, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Waterloo, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Hazard, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Rosedale, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Lansing, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, The Bronx, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Blue Ash, Ohio
  - Research Site, Easley, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Vancouver, Washington
- Australia (13):
  - Research Site, Bedford Park
  - Research Site, Bendigo
  - Research Site, Box Hill
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, Herston
  - Research Site, Kogarah
  - Research Site, Launceston
  - Research Site, Nedlands
  - Research Site, Port Macquarie
  - Research Site, Randwick
  - Research Site, Westmead
  - Research Site, Woolloongabba
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Gilly
  - Research Site, Leuven
  - Research Site, Libramont-Chevigny
  - Research Site, Liège
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Toronto
- Chile (2):
  - Research Site, Santiago
  - Research Site, Viña del Mar
- France (14):
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Brest
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Pau
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (8):
  - Research Site, Berlin
  - Research Site, Esslingen am Neckar
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Löwenstein
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Villingen-Schwenningen
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Miskolc
- Israel (2):
  - Research Site, Haifa
  - Research Site, Jerusalem
- Italy (8):
  - Research Site, Aviano
  - Research Site, Catania
  - Research Site, Cremona
  - Research Site, Lecce
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
- Japan (27):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Habikino-shi
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Ube-shi
  - Research Site, Yokohama
- Mexico (4):
  - Research Site, Cuautitlán Izcalli
  - Research Site, Monterrey
  - Research Site, Oaxaca City
  - Research Site, Orizaba
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Rotterdam
  - Research Site, Tilburg
- Research Site, Lima, Peru
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Lublin
  - Research Site, Warsaw
- Research Site, Singapore, Singapore
- Slovakia (4):
  - Research Site, Bardejov
  - Research Site, Košice
  - Research Site, Nové Zámky
  - Research Site, Trnava
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Pretoria
  - Research Site, Vereeniging
- South Korea (7):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Hwasun-gun
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Girona
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Muang
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Konya
  - Research Site, Malatya
- United Kingdom (3):
  - Research Site, Glasgow
  - Research Site, Manchester
  - Research Site, Truro
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Naidoo J, Antonia S, Wu YL, Cho BC, Thiyagarajah P, Mann H, Newton M, Faivre-Finn C. Brief Report: Durvalumab After Chemoradiotherapy in Unresectable Stage III EGFR-Mutant NSCLC: A Post Hoc Subgroup Analysis From PACIFIC. J Thorac Oncol. 2023 May;18(5):657-663. doi: 10.1016/j.jtho.2023.02.009. Epub 2023 Feb 24. PMID 36841540
- [Derived] Senan S, Ozguroglu M, Daniel D, Villegas A, Vicente D, Murakami S, Hui R, Faivre-Finn C, Paz-Ares L, Wu YL, Mann H, Dennis PA, Antonia SJ. Outcomes with durvalumab after chemoradiotherapy in stage IIIA-N2 non-small-cell lung cancer: an exploratory analysis from the PACIFIC trial. ESMO Open. 2022 Apr;7(2):100410. doi: 10.1016/j.esmoop.2022.100410. Epub 2022 Mar 2. PMID 35247871
- [Derived] Naidoo J, Vansteenkiste JF, Faivre-Finn C, Ozguroglu M, Murakami S, Hui R, Quantin X, Broadhurst H, Newton M, Thiyagarajah P, Antonia SJ. Characterizing immune-mediated adverse events with durvalumab in patients with unresectable stage III NSCLC: A post-hoc analysis of the PACIFIC trial. Lung Cancer. 2022 Apr;166:84-93. doi: 10.1016/j.lungcan.2022.02.003. Epub 2022 Feb 9. PMID 35245844
- [Derived] Spigel DR, Faivre-Finn C, Gray JE, Vicente D, Planchard D, Paz-Ares L, Vansteenkiste JF, Garassino MC, Hui R, Quantin X, Rimner A, Wu YL, Ozguroglu M, Lee KH, Kato T, de Wit M, Kurata T, Reck M, Cho BC, Senan S, Naidoo J, Mann H, Newton M, Thiyagarajah P, Antonia SJ. Five-Year Survival Outcomes From the PACIFIC Trial: Durvalumab After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Apr 20;40(12):1301-1311. doi: 10.1200/JCO.21.01308. Epub 2022 Feb 2. PMID 35108059
- [Derived] Ouwens M, Darilay A, Zhang Y, Mukhopadhyay P, Mann H, Ryan J, Dennis PA. Assessing the Influence of Subsequent Immunotherapy on Overall Survival in Patients with Unresectable Stage III Non-Small Cell Lung Cancer from the PACIFIC Study. Curr Ther Res Clin Exp. 2021 Aug 12;95:100640. doi: 10.1016/j.curtheres.2021.100640. eCollection 2021. PMID 34484473
- [Derived] Socinski MA, Ozguroglu M, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Gray JE, Park K, Vincent M, Mann H, Newton M, Dennis PA, Antonia SJ. Durvalumab After Concurrent Chemoradiotherapy in Elderly Patients With Unresectable Stage III Non-Small-Cell Lung Cancer (PACIFIC). Clin Lung Cancer. 2021 Nov;22(6):549-561. doi: 10.1016/j.cllc.2021.05.009. Epub 2021 Jun 12. PMID 34294595
- [Derived] Garassino MC, Paz-Ares L, Hui R, Faivre-Finn C, Spira A, Planchard D, Ozguroglu M, Daniel D, Vicente D, Murakami S, Langer C, Senan S, Spigel D, Ryden A, Zhang Y, O'Brien C, Dennis PA, Antonia SJ. Patient-reported outcomes with durvalumab by PD-L1 expression and prior chemoradiotherapy-related variables in unresectable stage III non-small-cell lung cancer. Future Oncol. 2021 Apr;17(10):1165-1184. doi: 10.2217/fon-2020-1102. Epub 2021 Feb 15. PMID 33583206
- [Derived] Mehra R, Yong C, Seal B, van Keep M, Raad A, Zhang Y. Cost-Effectiveness of Durvalumab After Chemoradiotherapy in Unresectable Stage III NSCLC: A US Healthcare Perspective. J Natl Compr Canc Netw. 2021 Feb 2;19(2):153-162. doi: 10.6004/jnccn.2020.7621. Print 2021 Feb. PMID 33545688
- [Derived] Faivre-Finn C, Vicente D, Kurata T, Planchard D, Paz-Ares L, Vansteenkiste JF, Spigel DR, Garassino MC, Reck M, Senan S, Naidoo J, Rimner A, Wu YL, Gray JE, Ozguroglu M, Lee KH, Cho BC, Kato T, de Wit M, Newton M, Wang L, Thiyagarajah P, Antonia SJ. Four-Year Survival With Durvalumab After Chemoradiotherapy in Stage III NSCLC-an Update From the PACIFIC Trial. J Thorac Oncol. 2021 May;16(5):860-867. doi: 10.1016/j.jtho.2020.12.015. Epub 2021 Jan 19. PMID 33476803
- [Derived] Faivre-Finn C, Spigel DR, Senan S, Langer C, Perez BA, Ozguroglu M, Daniel D, Villegas A, Vicente D, Hui R, Murakami S, Paz-Ares L, Broadhurst H, Wadsworth C, Dennis PA, Antonia SJ. Impact of prior chemoradiotherapy-related variables on outcomes with durvalumab in unresectable Stage III NSCLC (PACIFIC). Lung Cancer. 2021 Jan;151:30-38. doi: 10.1016/j.lungcan.2020.11.024. Epub 2020 Nov 26. PMID 33285469
- [Derived] Paz-Ares L, Spira A, Raben D, Planchard D, Cho BC, Ozguroglu M, Daniel D, Villegas A, Vicente D, Hui R, Murakami S, Spigel D, Senan S, Langer CJ, Perez BA, Boothman AM, Broadhurst H, Wadsworth C, Dennis PA, Antonia SJ, Faivre-Finn C. Outcomes with durvalumab by tumour PD-L1 expression in unresectable, stage III non-small-cell lung cancer in the PACIFIC trial. Ann Oncol. 2020 Jun;31(6):798-806. doi: 10.1016/j.annonc.2020.03.287. Epub 2020 Mar 21. PMID 32209338
- [Derived] Gray JE, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, Cho BC, Planchard D, Paz-Ares L, Faivre-Finn C, Vansteenkiste JF, Spigel DR, Wadsworth C, Taboada M, Dennis PA, Ozguroglu M, Antonia SJ. Three-Year Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC-Update from PACIFIC. J Thorac Oncol. 2020 Feb;15(2):288-293. doi: 10.1016/j.jtho.2019.10.002. Epub 2019 Oct 14. PMID 31622733
- [Derived] Hui R, Ozguroglu M, Villegas A, Daniel D, Vicente D, Murakami S, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Gray JE, Ryden A, Viviers L, Poole L, Zhang Y, Dennis PA, Antonia SJ. Patient-reported outcomes with durvalumab after chemoradiotherapy in stage III, unresectable non-small-cell lung cancer (PACIFIC): a randomised, controlled, phase 3 study. Lancet Oncol. 2019 Dec;20(12):1670-1680. doi: 10.1016/S1470-2045(19)30519-4. Epub 2019 Oct 7. PMID 31601496
- [Derived] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Derived] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- See also: AstraZeneca Cancer Study Locator Service astrazeneca@emergingmed.com 1-877-400-465 — http://www.emergingmed.com/networks/AstraZeneca
- See also: CSR redacted synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191C00001&attachmentIdentifier=5253288a-15c6-48e2-a5b4-20315b70234e&fileName=D4191C00001-CSR_synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized between 09 May 2014 and 22 Apr 2016 in 235 study centers across 26 countries. Data cut-off (DCO) date for analysis of progression-free survival (PFS) and PFS rates at 12 and 18 months: 13 Feb 2017; DCO date for analysis of overall survival (OS) and all other secondary outcome measures: 22 Mar 2018; DCO date for completion of long-term survival: 11 Jan 2021.
Pre-assignment Details: Eligible patients with locally advanced, unresectable Stage III non-small cell lung cancer were randomized in a 2:1 ratio to receive either durvalumab (MEDI4736) 10 milligrams (mg) / kilogram (kg) every 2 weeks (Q2W) or placebo.
Groups:
- Durvalumab (MEDI4736): Patients in the durvalumab (MEDI4736) monotherapy group were to receive durvalumab 10 mg/kg Q2W via intravenous infusion for up to 12 months.
- Placebo: Patients in the placebo group were to receive matching placebo for intravenous infusion Q2W for up to 12 months.
Period: Overall Study
Arm/Group | Durvalumab (MEDI4736) | Placebo
Started (Randomized) | 476 | 237
Full Analysis Set (FAS) | 476 | 237
Received Treatment | 473 | 236
Safety Analysis Set | 475 | 234
Completed 12 Months of Treatment | 232 | 82
Completed (Ongoing study at final DCO (study complete)) | 178 | 68
Not Completed | 298 | 169
Not completed — Withdrawal by Subject | 30 | 16
Not completed — Lost to Follow-up | 8 | 3
Not completed — Death | 260 | 149
Not completed — Missing Termination Reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on the FAS consisting of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab (MEDI4736) | Placebo | Total
Number analyzed (Participants) | 476 | 237 | 713
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.66) | 62.6 (9.64) | 62.9 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 71 | 213
  Male | 334 | 166 | 500
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 337 | 157 | 494
  Black or African American | 12 | 2 | 14
  Asian | 120 | 72 | 192
  Native Hawaiian or Pacific Islander | 1 | 1 | 2
  American Indian or Alaska Native | 4 | 5 | 9
  Other | 1 | 0 | 1
  Missing | 1 | 0 | 1
Smoking History [Count of Participants; unit: Participants]
  Non-smoker | 43 | 21 | 64
  Ex-smoker | 354 | 178 | 532
  Current smoker | 79 | 38 | 117

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Based on Blinded Independent Central Review (BICR) According to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: PFS was defined as the time from randomization until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression). Progression was defined using RECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed until 13 Feb 2017 DCO; up to a maximum of approximately 3 years.
Population: FAS included all randomized patients, analyzed on an intent-to-treat (ITT) basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Months | 16.8 [13.0 to 18.1] | 5.6 [4.6 to 7.8]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; Analysis performed using a stratified log rank test adjusting for age at randomization (<65 vs ≥65), sex (male vs female), and smoking history (smoker vs non-smoker) with ties handled using the Breslow approach; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.42 to 0.65]

2. Primary Outcome: Overall Survival
Description: OS was defined as the time from the date of randomization until death due to any cause. OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline until death due to any cause. Assessed until 22 Mar 2018 DCO; up to a maximum of approximately 4 years.
Population: FAS included all randomized patients, analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Months | NA [34.7 to NA] — The median and upper limit of 95% confidence interval (CI) could not be calculated as they were not reached. | 28.7 [22.9 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.00251, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.53 to 0.87]

3. Secondary Outcome: Objective Response Rate (ORR) Based on BICR Assesments According to RECIST 1.1
Description: ORR was defined as the percentage of patients with at least one visit response of Complete Response (CR) or Partial Response (PR) per RECIST 1.1 for target lesions: CR: Disappearance of all target lesions; PR: >=30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR.
Time Frame: Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~ 12 weeks thereafter until confirmed disease progression. Assessed until 22 Mar 2018 DCO; up to a maximum of approximately 4 years.
Population: FAS (which included all randomized patients) with measureable disease at baseline, analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 443 | 213
Percentage of patients | 30.0 [25.79 to 34.53] | 17.8 [12.95 to 23.65]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; Analysis performed using Fisher's exact test with mid p-value modification by subtracting half of the probability of the observed table from Fisher's p-value; Test type: Superiority; p < 0.001, Fisher Exact

4. Secondary Outcome: Duration of Response (DoR) Based on BICR Assessments According to RECIST 1.1
Description: DoR was defined as the time from date for first documented response of CR or PR until the first documented response of progression per RECIST 1.1 or death in the absence of progression. DoR was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 3
Population: FAS included all randomized patients, analyzed on an ITT basis. Only patients with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 133 | 38
Months | NA [27.4 to NA] — The median and upper limit of 95% CI could not be calculated as they were not reached. | 18.4 [6.7 to 24.5]

5. Secondary Outcome: Proportion of Patients Alive and Progression Free at 12 Months From (APF12) Based on BICR Assessments According to RECIST 1.1
Description: APF12 was defined as the percentage of patients who were alive and progression free per RECIST 1.1 at 12 months after randomization per Kaplan-Meier estimate of PFS at 12 months.
Time Frame: Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~ 12 weeks thereafter until confirmed disease progression. Assessed until 13 Feb 2017 DCO; up to a maximum of approximately 3 years.
Population: FAS included all randomized patients, analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Percentage of patients | 55.9 [51.0 to 60.4] | 35.3 [29.0 to 41.7]

6. Secondary Outcome: Proportion of Patients Alive and Progression Free at 18 Months From (APF18) Based on BICR Assessments According to RECIST 1.1
Description: APF18 was defined as the percentage of patients who were alive and progression free per RECIST 1.1 at 18 months after randomization per the Kaplan-Meier estimate of PFS at 18 months.
Time Frame: as for outcome 5
Population: FAS included all randomized patients, analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Percentage of patients | 44.2 [37.7 to 50.5] | 27.0 [19.9 to 34.5]

7. Secondary Outcome: Time to Death or Distant Metastasis (TTDM) Based on BICR Assessments According to RECIST 1.1
Description: TTDM was defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis. Distant metastasis was defined as any new lesion that was outside of the radiation field according to RECIST 1.1 or proven by biopsy. TTDM was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 3
Population: FAS included all randomized patients, analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Months | 28.3 [24.0 to 34.9] | 16.2 [12.5 to 21.1]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.41 to 0.68]

8. Secondary Outcome: Percentage of Patients Alive at 24 Months (OS24)
Description: OS24 was defined as the percentage of patients who were alive at 24 months after randomization per the Kaplan-Meier estimate of OS at 24 months.
Time Frame: From baseline until death due to any cause. Assessed until 22 Mar 2018 DCO; up to a maximum of approximately 4 years.
Population: FAS included all randomized patients, analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Percentage of patients | 66.3 [61.7 to 70.4] | 55.6 [48.9 to 61.8]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; Test type: Superiority; p = 0.005, z-test — P-value generated based on z-test where z-test statistic is the ratio of the log-transformed ratio of the cumulative hazards in the 2 treatment arms divided by the square root of the variance; The variance was estimated using the delta method and Greenwood's formula

9. Secondary Outcome: Time to Second Progression or Death (PFS2)
Description: PFS2 was defined as the time from randomization to the time of the second progression or death. The date of second progression was recorded by the investigator and defined according to local standard clinical practice, and could have involved any of the following: objective radiological, symptomatic progression, or death. RECIST assessments were not collected for assessment of PFS2. PFS2 was calculated using the Kaplan-Meier technique.
Time Frame: Following confirmed progression, patients were assessed every ~12 weeks until second disease progression. Assessed until 22 Mar 2018 DCO; up to a maximum of approximately 4 years.
Population: FAS included all randomized patients, analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Months | 28.3 [25.1 to 34.7] | 17.1 [14.5 to 20.7]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.46 to 0.73]

10. Secondary Outcome: Time to Deterioration of Global Health Status / Health-Related Quality of Life (HRQoL), Assessed Using European Organization for Research and Treatment of Cancer 30-Item Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Global health status/HRQoL was assessed using the EORTC QLQ-C30 global QoL scale which includes 2 items from the QLQ-C30: "How would you rate your overall health during the past week?" (Item 29) and "How would you rate your overall QoL during the past week?" (Item 30). Scores from 0 to 100 were derived for each item with higher scores indicating a better health status. Time to deterioration for global health status/HRQoL was defined as time from randomization until the date of first clinically meaningful deterioration (a decrease in global health status/HRQoL from baseline of ≥10) or death (by any cause) in the absence of a clinically meaningful deterioration. Time to deterioration was calculated using the Kaplan-Meier technique.
Time Frame: At baseline, every 4 weeks for first 8 weeks, then every ~8 weeks until 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed until 22 Mar 2018 DCO; up to a maximum of approximately 4 years.
Population: FAS included all randomized patients, analyzed on an ITT basis. Only patients with baseline scores ≥ 10 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Months | 7.4 [5.5 to 9.3] | 5.7 [4.2 to 10.5]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; The hazard ratio and CI were estimated from a stratified Cox proportional hazards model with the Breslow method to control for ties, the stratification factors age at randomization (<65 vs ≥65), sex (male vs female) and smoking history (smoker vs non-smoker) in the strata statement, and the CI calculated using a profile likelihood approach; Test type: Superiority; p = 0.664, Log Rank — Analysis performed using a stratified log rank test adjusting for age at randomization (<65 vs ≥65), sex (male vs female), and smoking history (smoker vs non-smoker) with ties handled using the Breslow approach; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.77 to 1.18]

11. Secondary Outcome: Time to Deterioration of Primary Patient-Reported Outcome (PRO) Symptoms, Assessed Using European Organization for Research and Treatment of Cancer QoL Lung Cancer Module (EORTC QLQ-LC13)
Description: The EORTC QLQ-LC13 is a lung cancer specific module from the EORTC comprising 13 questions to assess lung cancer symptoms (cough, hemoptysis, dyspnea, chest pain, arm/shoulder pain, and other pain), treatment related side-effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication. Scores from 0 to 100 were derived for each symptom item with higher scores representing greater symptom severity. Time to symptom deterioration was defined as time from randomization until the date of first clinically meaningful symptom deterioration (an increase in the score from baseline of ≥10) or death (by any cause) in the absence of a clinically meaningful symptom deterioration. Results are presented for time to deterioration in the following PRO endpoints identified as primary for EORTC QLQ-LC13: dyspnea, cough, hemoptysis and chest pain. Time to deterioration was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 10
Population: FAS included all randomized patients, analyzed on an ITT basis. Only patients with baseline scores ≤ 90 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 476 | 237
Months
  Dyspnea: number analyzed (Participants) | 467 | 230
  Dyspnea | 2.8 [1.9 to 3.7] | 3.7 [2.3 to 4.1]
  Cough: number analyzed (Participants) | 442 | 216
  Cough | 5.6 [4.5 to 7.3] | 5.6 [3.7 to 6.0]
  Hemoptysis: number analyzed (Participants) | 472 | 232
  Hemoptysis | NA [NA to NA] — The median and 95% CIs could not be calculated as they were not reached. | 29.6 [21.2 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  Chest pain: number analyzed (Participants) | 463 | 229
  Chest pain | 11.1 [7.4 to 18.6] | 8.3 [5.6 to 13.8]
Statistical Analysis 1: Comparison: Durvalumab (MEDI4736) vs Placebo; Treatment comparison for dyspnea. The hazard ratio and CI were estimated from a stratified Cox proportional hazards model with the Breslow method to control for ties, the stratification factors age at randomization (<65 vs ≥65), sex (male vs female) and smoking history (smoker vs non-smoker) in the strata statement, and the CI calculated using a profile likelihood approach; Test type: Superiority; p = 0.522, Log Rank — [p-value comment as in outcome 10, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.88 to 1.29]
Statistical Analysis 2: Comparison: Durvalumab (MEDI4736) vs Placebo; Treatment comparison for cough. The hazard ratio and CI were estimated from a stratified Cox proportional hazards model with the Breslow method to control for ties, the stratification factors age at randomization (<65 vs ≥65), sex (male vs female) and smoking history (smoker vs non-smoker) in the strata statement, and the CI calculated using a profile likelihood approach; Test type: Superiority; p = 0.380, Log Rank — [p-value comment as in outcome 10, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.12]
Statistical Analysis 3: Comparison: Durvalumab (MEDI4736) vs Placebo; Treatment comparison for hemoptysis. The hazard ratio and CI were estimated from a stratified Cox proportional hazards model with the Breslow method to control for ties, the stratification factors age at randomization (<65 vs ≥65), sex (male vs female) and smoking history (smoker vs non-smoker) in the strata statement, and the CI calculated using a profile likelihood approach; Test type: Superiority; p = 0.048, Log Rank — [p-value comment as in outcome 10, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.56 to 1.00]
Statistical Analysis 4: Comparison: Durvalumab (MEDI4736) vs Placebo; Treatment comparison for chest pain. The hazard ratio and CI were estimated from a stratified Cox proportional hazards model with the Breslow method to control for ties, the stratification factors age at randomization (<65 vs ≥65), sex (male vs female) and smoking history (smoker vs non-smoker) in the strata statement, and the CI calculated using a profile likelihood approach; Test type: Superiority; p = 0.626, Log Rank — [p-value comment as in outcome 10, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.19]

12. Secondary Outcome: Pharmacokinetics (PK) of Durvalumab; Peak and Trough Serum Concentrations
Description: To evaluate PK, blood samples were collected pre-dose and post-dose and trough and peak serum concentrations of durvalumab, respectively, were determined. Pre-dose samples were taken within 60 minutes before infusion and post-dose samples were taken within 10 minutes after the end of infusion.
Time Frame: Samples were collected pre-dose on Day 1 (Week 0), Week 8, Week 24 and Week 48, and post-dose on Day 1 (Week 0) and Week 24. Analysis performed at 22 Mar 2018 DCO.
Population: PK analysis set included all patients who received at least 1 dose of durvalumab per the protocol, for whom any post-dose data were available, and who did not violate or deviate from the protocol in ways that would significantly affect the PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Durvalumab (MEDI4736)
Number analyzed (Participants) | 473
Micrograms per milliliter
  Week 0: peak concentration: number analyzed (Participants) | 385
  Week 0: peak concentration | 191.00 (72.4)
  Week 8: trough concentration: number analyzed (Participants) | 289
  Week 8: trough concentration | 120.00 (62.2)
  Week 24: trough concentration: number analyzed (Participants) | 225
  Week 24: trough concentration | 177.00 (47.9)
  Week 24: peak concentration: number analyzed (Participants) | 207
  Week 24: peak concentration | 373.00 (43.6)
  Week 48: trough concentration: number analyzed (Participants) | 213
  Week 48: trough concentration | 186.00 (67.4)

13. Secondary Outcome: Number of Patients With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: ADA positive post-baseline only was also referred to as treatment-induced ADA positive. Treatment-boosted ADA was defined as baseline positive ADA titer that was boosted by ≥4-fold following drug administration. Persistently positive was defined as positive at ≥2 post-baseline assessments (with ≥16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Confirmed ADA positive samples were subsequently tested in a neutralizing antibody assay.
Time Frame: Samples were collected pre-dose on Day 1 (Week 0), Week 8, Week 24 and Week 48. Analysis performed at 22 Mar 2018 DCO.
Population: ADA evaluable population included patients who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA results.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab (MEDI4736) | Placebo
Number analyzed (Participants) | 416 | 204
Participants
  ADA positive at any visit | 19 | 10
  ADA positive post-baseline only | 8 | 5
  Treatment-boosted ADA positive | 0 | 0
  ADA positive at baseline and post-baseline | 2 | 2
  ADA positive at baseline only | 9 | 3
  ADA persistently positive | 5 | 5
  ADA transient positive | 5 | 2
  Neutralizing antibodies positive at any visit | 3 | 0

ADVERSE EVENTS:
Time Frame: Serious and Other (non-serious) treatment-emergent adverse event (TEAE) data collected during the 12-month treatment period. All-cause mortality (death due to any cause) collected for entire duration of the study. Assessed until 11 Jan 2021 DCO for completion of long-term survival; approximately 5 years from last patient enrolled.
Description: TEAEs included events from first dose of study drug until the earlier of 90 days after last dose or date of first subsequent therapy. 473 and 236 patients in the durvalumab and placebo groups, respectively, received treatment but 2 patients randomized to placebo received 1 dose of durvalumab in error and are included in the durvalumab safety analysis set.
Arm/Group | Durvalumab (MEDI4736) | Placebo
All-Cause Mortality (participants affected / at risk) | 262/475 | 154/234
Serious Adverse Events (participants affected / at risk) | 138/475 | 54/234
Other Adverse Events (participants affected / at risk) | 436/475 | 212/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (MEDI4736) (N=475) | Placebo (N=234)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (7) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Eosinophilic myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 33 (39) | 14 (16)
Pneumonia adenoviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
West Nile viral infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (5) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 7 (8)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Endotoxaemia (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 2 (3)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 17 (17) | 4 (5)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus prostatic (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (MEDI4736) (N=475) | Placebo (N=234)
Anaemia (Blood and lymphatic system disorders) | 35 (39) | 26 (32)
Hyperthyroidism (Endocrine disorders) | 35 (39) | 4 (4)
Hypothyroidism (Endocrine disorders) | 54 (62) | 4 (4)
Constipation (Gastrointestinal disorders) | 57 (59) | 20 (27)
Diarrhoea (Gastrointestinal disorders) | 87 (136) | 46 (56)
Vomiting (Gastrointestinal disorders) | 36 (45) | 19 (25)
Upper respiratory tract infection (Infections and infestations) | 57 (69) | 24 (30)
Nausea (Gastrointestinal disorders) | 68 (88) | 31 (43)
Asthenia (General disorders) | 51 (73) | 31 (50)
Fatigue (General disorders) | 114 (130) | 47 (52)
Urinary tract infection (Infections and infestations) | 28 (42) | 13 (13)
Dizziness (Nervous system disorders) | 33 (36) | 22 (25)
Headache (Nervous system disorders) | 52 (58) | 21 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 169 (220) | 59 (75)
Non-cardiac chest pain (General disorders) | 35 (39) | 21 (22)
Oedema peripheral (General disorders) | 37 (41) | 9 (10)
Pyrexia (General disorders) | 70 (92) | 22 (23)
Bronchitis (Infections and infestations) | 33 (44) | 19 (22)
Nasopharyngitis (Infections and infestations) | 42 (51) | 14 (18)
Pneumonia (Infections and infestations) | 48 (54) | 12 (14)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 80 (84) | 33 (33)
Decreased appetite (Metabolism and nutrition disorders) | 69 (84) | 29 (32)
Hypokalaemia (Metabolism and nutrition disorders) | 24 (33) | 12 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 83 (110) | 44 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 50 (55) | 27 (31)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 25 (27) | 18 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (41) | 10 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (35) | 14 (14)
Paraesthesia (Nervous system disorders) | 22 (24) | 12 (13)
Insomnia (Psychiatric disorders) | 45 (47) | 17 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 106 (133) | 57 (67)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 44 (46) | 11 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 46 (53) | 19 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 37 (38) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 60 (70) | 14 (17)
Rash (Skin and subcutaneous tissue disorders) | 61 (72) | 18 (23)
Hypertension (Vascular disorders) | 26 (29) | 8 (8)

LIMITATIONS AND CAVEATS:
Results of interim PFS analysis are considered as final PFS analysis; results of interim OS analysis are considered as final OS analysis. Patients were followed up for long-term survival until approximately 5 years after last patient enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT02125461/Prot_004.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02125461/SAP_005.pdf